CLINICAL TRIAL: NCT07128862
Title: Effects of Heavy-load Resistance Training With and Without Blood Flow Restriction Therapy on Quadriceps Muscle Strength and Endurance in Athletes
Brief Title: Heavy-load Resistance Training With and Without Blood Flow Restriction Therapy in Athletes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0461
Record Dates: First submitted 2025-07-21; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Sports Physical Therapy

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial
Who Masked: Outcomes Assessor
Masking Description: Assesor Blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Heavy-Load Resistance Training with Blood Flow Restriction (Experimental): In this group, the participants will perform three important exercises namely back squats, leg press, and bench press. Those exercises were performed at a training intensity ranging from 70-80% of each person's 1-repetition maximum (1RM). 12 cm pneumatic cuffs was placed proximally on the thigh (for exercise of lower body) and arm (for exercise of upper body), and blood flow restriction was applied through them. Doppler ultrasound was used weekly to measure limb occlusion pressure (LOP) to then set the cuff pressure at 50% of each participant's predetermined LOP. During working sets it was made the cuffs inflated but during rest periods they were deflated. The exercise protocol consists of:
  Interventions: Other: Heavy-Load Resistance Training with Blood Flow Restriction
- Heavy-Load Resistance Training Only (HLRT) (Experimental): This control group will perform the identical exercise protocol (same exercises, intensities, volumes, and rest periods) as the BFR group, but without any blood flow restriction application. The same progression criteria will be used for both groups to ensure comparable training stimulus.
  Interventions: Other: Heavy-Load Resistance Training Only

INTERVENTIONS:
Other: Heavy-Load Resistance Training with Blood Flow Restriction — Blood Flow Restriction (BFR) Training (also known as "Kaatsu" training is an innovative and increasingly popular exercise technique to improve muscle strength and hypertrophy with relatively low loads. Heavy Load Resistance Training (HL-RT) is one of the most effective exercise methodology that is widely used to increase muscular strength and hypertrophy.
  Arms: Heavy-Load Resistance Training with Blood Flow Restriction
Other: Heavy-Load Resistance Training Only — Heavy Load Resistance Training (HL-RT) is one of the most effective exercise methodology that is widely used to increase muscular strength and hypertrophy.
  Arms: Heavy-Load Resistance Training Only (HLRT)

SUMMARY:
A 8 weeks, single-blinded randomized controlled trial will be conducted at Pakistan Sports Board (PSB). Forty-four athletes (18-35 years) will be randomized into Group A (HL-RT + BFR, n = 22) and Group B (HL-RT only, n = 22). BFR will be applied at 50% limb occlusion pressure during lower-body exercises (squats, leg press). Both groups trained 3x/week for 4 weeks at 70-80% 1RM. Outcomes included 1RM strength, squat endurance, push-up performance, and International Physical Activity Questionnaire (IPAQ) scores.

DETAILED DESCRIPTION:
This study is a single-blinded randomized controlled trial (RCT) comparing heavy-load resistance training (HLRT) with blood flow restriction (BFR) versus HLRT alone. Participants will be blinded to group allocation, but outcome assessors will not remain blinded throughout the study.

Group A participants will perform three important exercises namely back squats, leg press, and bench press. Those exercises were performed at a training intensity ranging from 70-80% of each person's 1-repetition maximum (1RM). 12 cm pneumatic cuffs was placed proximally on the thigh (for exercise of lower body) and arm (for exercise of upper body), and blood flow restriction was applied through them. Doppler ultrasound was used weekly to measure limb occlusion pressure (LOP) to then set the cuff pressure at 50% of each participant's predetermined LOP. During working sets it was made the cuffs inflated but during rest periods they were deflated. The exercise protocol consists of:

* Back squats: 4 sets of 6 repetitions
* Leg press: 3 sets of 8 repetitions
* Bench press: 3 sets of 10 repetitions All sets will be followed by a standardized 2-minute rest period. Training load will progressively increased by 2.5-5% when participants can complete all prescribed repetitions with proper form for two consecutive sessions.

Group B: Heavy-Load Resistance Training Only (HLRT) This control group will perform the identical exercise protocol (same exercises, intensities, volumes, and rest periods) as the BFR group, but without any blood flow restriction application. The same progression criteria will be used for both groups to ensure comparable training stimulus.

Post-Intervention Data Collection (Week 4)

Following the 4-week intervention period, all participants were undergone reassessment using the same measures collected at baseline:

1. 1RM testing for back squat and bench press
2. Muscular endurance tests (max repetition squat test and 1-minute push-up test)
3. International Physical Activity Questionnaire (IPAQ)

ELIGIBILITY:
Inclusion Criteria:

* Participants with age between 18 and 35 years.
* Active individual participating in sport activities at least 3 times a week for the past 6 months.
* Participants with any non-heart conditions.
* Individuals voluntarily participating and providing informed consent.
* Sprinters, Footballer

Exclusion Criteria:

* Individuals with DVT or other pulmonary artery disease.
* Pregnant women or those planning to become pregnant.
* Participants with recent musculoskeletal injuries (within the 6 months).
* Individuals currently involved in another study.
* Participants allergic to or sensitive to the materials used in the BFR bands.
* Individuals who anticipate being unable to attend all training sessions.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-07-30 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-09-02 (Estimated)

PRIMARY OUTCOMES:
1RM strength | 6 weeks
  The 1 Repetition Maximum (1 RM) Testing protocol determines quadriceps maximal strength through identifying the maximum weight an individual can lift in a single attempt with exercises that include the leg press or squat and leg extension movements.
Squat Endurance | 6 weeks
  Experts have established the validity of 3-5 RM squats as a strength test because they correlate strongly with quadriceps force output and exhibit excellent reliability (ICC > 0.90) through standardization of stance and depth and rest periods. Maximal bodyweight squats at 60-70% 1 RM or to complete failure serve as reliable (ICC ~0.70-0.85) and moderate tests of endurance even though hip and core involvement affects validity.
Push Up Performance | 6 weeks
  The push-up test is largely used to evaluate upper body endurance and strength (chest, shoulders, triceps) without much activation of the quadriceps and should not be considered as an indicator of quad endurance or strength. On standard push ups though, quads serve only as stabilizers which means it does not provide much of contribution than exercise such as squatting or doing leg extensions. Push-ups can still be considered a reliable test (ICC ~0.80-0.90) for upper body muscular endurance but cannot be used to assess quadriceps function
International Physical Activity Questionnaire (IPAQ) scores | 6 weeks
  International Physical Activity Questionnaire (IPAQ). Interpretation: Higher score indicates increased physical activity in athletes. Effect of interpretation: BFR with heavy load training significantly increases physical activity levels as compared to control.
  Description: The International Physical Activity Questionnaire - short form (IPAQ-SF) will be used to assess a participant's total physical activity levels. This self-report tool estimates MET-minutes per week across various domains. The score ranges from 0 to an upper limit, with higher scores indicating greater levels of physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Hassan, MSPT, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Sports Board, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No